CLINICAL TRIAL: NCT05247411
Title: Nurse Educational Intervention Improves Symptoms Control and Compliance in Fibromyalgia Patients on Medical Cannabis Therapy
Brief Title: Nurse Educational Intervention to Improve Symptoms in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Antonio Biagio Torsello, Professor, University of Milano Bicocca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Education and Fibromyalgia 545
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; nurse; nursing; medical cannabis; education; interview
MeSH Terms: conditions — Fibromyalgia | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational intervention (Experimental): a Skype-videoconference, which included a 30 min educational intervention, was held with each subject.
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — During the videoconference, the following items were investigated and evaluated:
  (i) Knowledge on FM: knowledge on symptoms, onset, treatment, strategies and non-pharmacological interventions that can be implemented to improve the quality of life (physical exercise, nutrition, participation in meditative movement practices, mutual aid groups, membership in a patient association, etc.); (ii) Any MC intake or interest in starting the intake of MC; (iii) Knowledge on MC therapy: specific knowledge on the drug, correct intake, adherence, treatment of side effects related to intake and strategies to reduce them; (iv) Self-care: how the person manages his personal life despite a chronic disease, how she or he monitors, recognizes and treats the symptoms in terms of timing and quality; possible presence of caregivers in their life who help in the management of the disease; employment and how FM affects it and daily life.

SUMMARY:
To improve self-care and therapy adherence by fibromyalgia (FM) patients through a nursing educational intervention. Historic diagnoses of subjects included terms such as "insane", "imaginary ill", "whiny"; as well, their physical conditions were underestimated by their immediate families. All subjects have problematic employment histories which consistently identified their varied employments as physically too demanding. Over time, increased physician- and societal-awareness, resulted in all subjects being diagnosed with FM; consequently, all subjects reported a strong desire to become well-informed about FM and its treatment. Although medical cannabis (MC) was an available therapy, twenty subjects reported that cannabis had never been proposed despite years of ineffective therapies. In this tudy the effects of a educational intervention by expert nurses on fibromyalgia and MC use were investigated.

DETAILED DESCRIPTION:
Aims This study aims to evaluate the knowledge of fibromyalgia patients who use therapeutic cannabis or are interested in taking it, introducing the figure of the nurse in the therapeutic path of patients. The primary objective was to increase the knowledge relating to FM (in terms of symptoms, onset, treatment strategies that can improve the quality of life), self-care and adherence through a nursing educational intervention. The secondary objective was to evaluate the efficacy of the nursing educational intervention, using validated clinimetric scales.

Design We performed a qualitative study with face-to-face semi-structured interviews and patient tailored educational interventions. Two weeks before the interview, subjects were asked to complete the Fibromyalgia Impact Questionnaire Revised (FIQR) and the A-14 Scale online. Two weeks after the interview, patients were asked to complete the same questionnaires in addition the Clinical Global Impression - Global Improvement (CGI-I) Scale. This study adheres to the Consolidated criteria for Reporting Qualitative research (COREQ).

Data collection After obtaining written informed consent for participation in the study, each participant was asked to complete online the Fibromyalgia Impact Questionnaire Revised (FIQR) and The A-14 Scale. Two weeks after completing these online questionnaires, a Skype-videoconference, which included a 30 min educational intervention, was held with each subject. Two weeks after the videoconference, patients were required to complete the FIQR, The A-14 Scale, as well as the Clinical Global Impression - Global Improvement (CGI-I) Scale Data analysis Descriptive analyses were performed on study participants.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibromyalgia syndrome carried out for more than 3 months and confirmed by the specialist (rheumatologist / algologist);
* age> 18 years;
* ability to understand the objectives and methods of the study and to read and sign the informed consent form.

Exclusion Criteria:

• patients not in Medical Cannabis therapy and/or not interested in starting the therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Subjective improvement assessed with Fibromyalgia Impact Questionnaire Revised (FIQR) questionnaire | baseline and 14 days
  At baseline and two weeks after the videoconference, patients were required to complete the Fibromyalgia Impact Questionnaire Revised (FIQR), in order to assess effects of the educational intervention on therapeutic perspective and compliance. The FIQR is made of 21 items and the answers range between 0 (best performance) and 10 (worst performance)
Subjective improvement assessed with the A-14 Scale | baseline and 14 days
  At baseline and two weeks after the videoconference, patients were required to complete the A-14 Scale, in order to assess effects of the educational intervention on therapeutic perspective and compliance. The A-14 Scale is made up of 14 questions, which can be answered using a 5-element Likert-scale (from "never" [5] to "very often" [0]). The result of the scale ranges from "non-compliant" (score <50) to "compliant" (score 50-56)
Subjective improvement assessed with the Clinical Global Impression - Global Improvement (CGI-I) Scale | 14 days
  At two weeks after the videoconference, patients were required to complete the Clinical Global Impression - Global Improvement (CGI-I) Scale, which measures the subjective progress of the patient, in order to assess effects of the educational intervention on therapeutic perspective and compliance. Scores are the followings: 1 Minimally improved: 2 Much improved; 3 Very much improved; 4 No change; 5 Minimally worse; 6 Much worse; 7 Very much worse

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine, University of Milano-Bicocca, Monza, Italy

REFERENCES:
- [Result] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Result] Bennett RM, Friend R, Jones KD, Ward R, Han BK, Ross RL. The Revised Fibromyalgia Impact Questionnaire (FIQR): validation and psychometric properties. Arthritis Res Ther. 2009;11(4):R120. doi: 10.1186/ar2783. Epub 2009 Aug 10. PMID 19664287
- [Result] Jank S, Bertsche T, Schellberg D, Herzog W, Haefeli WE. The A14-scale: development and evaluation of a questionnaire for assessment of adherence and individual barriers. Pharm World Sci. 2009 Aug;31(4):426-431. doi: 10.1007/s11096-009-9296-x. Epub 2009 Apr 21. PMID 19381860
- [Result] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937